CLINICAL TRIAL: NCT01935843
Title: Clinical Study of Chimeric HER-2 Antigen Receptor-modified T Cells in Chemotherapy Refractory HER-2 Advanced Solid Tumors
Brief Title: Treatment of Chemotherapy Refractory Human Epidermalgrowth Factor Receptor-2( HER-2) Positive Advanced Solid Tumors
Acronym: CART-HER-2
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Professor and Director, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-009
Record Dates: First submitted 2013-09-01; First posted 2013-09-05 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Advanced HER-2 Positive Solid Tumors; Chemotherapy Refactory; HER-2 Antibody Inhibitor Therapy Refactory
Keywords: CART-HER-2; HER-2 positive; Advanced; Refactory; Solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anti-tumor responses of CART-HER-2 (Experimental)
  Interventions: Biological: CART-HER-2

INTERVENTIONS:
Biological: CART-HER-2

SUMMARY:
RATINALE: Placing a tumor antigen chimeric receptor that has been created in the laboratory into patient autologous T cells may make the body build immune response to kill cancer cells.

PURPOSE: This clinical trial is to study genetically engineered lymphocyte therapy in treating patients with HER-2 positive advanced solid tumors,such as breast cancer, gastric cancer, hepatic carcinoma, endometrial cancer and ovary cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I.Determine the safety and feasibility of the chimeric antigen receptor T cells transduced with anti-HER-2 vector(referred to as CART-HER-2 cells).

II.Determine duration of in vivo survival of CART-HER-2 cells. RT-PCR(reverse transcription polymerase chain reaction)analysis of whole blood will be used to detect and quantify survival of CART-HER-2 TCR zeta:CD137 and TCR(T-cell receptor) zeta cells over time.

SECONDARY OBJECTIVES:

I.For patients with detectable diseases, measure anti-tumor response due to CART-HER-2 cell infusions.

II.Estimate relative trafficking of CART-HER-2 cells in tumor bed.

III.Determine if cellular or humoral host immunity develops against the murine anti-HER-2, and assess correlation with loss of detectable CART-HER-2(loss of engraftment).

IV.Determine the relative subsets of CART-HER-2 T cells (Tcm,Tem,and Treg).

OUTLINE: Patients are assigned to 1 group according to order of enrollment. Patients receive anti-HER-2-CAR (coupled with CD137 and CD3 zeta signalling domains)vector-transduced autologous T cells on days 0,1, and 2 in the absence of unacceptable toxicity.

After completion of study treatment, patients are followed intensively for 6 months, every 3 months for 2 years, and annually thereafter for 13 years.

Estimate relative trafficking of CART-HER-2 cells in peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* Chemotherapy refractory HER-2-positive breast cancer, gastric cancer, non-small cell lung cancer, and chemotherapy resistant or relapsed ovary cancer.
* Relapsed patients after anti-HER-2 using antibody or kinase inhibitor therapy.
* Patients must be 18 years of age or older.
* Patients must have an ECOG (Eastern Cooperative Oncology Group )performance status of 0-2.
* Patients must have evidence of adequate bone marrow reserve, hepatic and renal function as evidenced by the following laboratory parameters:

Absolute neutrophil count greater than 1500/mm3. Platelet count greater than 100,000/mm3. Hemoglobin greater than 10g/dl (patients may receive transfusions to meet this parameter).

Total bilirubin < 1.5 times upper limits of normal. Serum creatinine less than or equal to 1.6 mg/ml or the creatinine clearance must be greater than 70 ml/min/1.73m(2).

* Seronegative for HIV antibody.
* Seronegative for active hepatitis B, and seronegative for hepatitis C antibody.
* Patients must be willing to practice birth control during and for four months following treatment.NOTE:women of child-bearing age must have evidence of negative pregnancy test.
* Patients must be willing to sign an informed consent.

Exclusion Criteria:

* Patients with life expectancy less than 12 months will be excluded.
* Patients with uncontrolled hypertension (> 160/95), unstable coronary disease evidenced by uncontrolled arrhythmias, unstable angina, decompensated congestive heart failure (> New York Heart Association Class II), or myocardial infarction within 6 months of study will be excluded.
* Patients with any of the following pulmonary function abnormalities will be excluded: FEV(forced expiratory volume), < 30% predicted; DLCO (diffusing capacity of lung for carbon monoxide) < 30% predicted (post-bronchodilator); Oxygen Saturation less than 90% on room air.
* Patients with severe liver and kidney dysfunction or consciousness disorders will be excluded.
* Pregnant and/or lactating women will be excluded.
* Patients with active infections, including HIV, will be excluded, due to unknown effects of the vaccine on lymphoid precursors.
* Patients with any type of primary immunodeficiencies will be excluded from the study.
* Patients requiring corticosteroids (other than inhaled) will be excluded.
* Patients with history of T cell tumors will be excluded.
* Patients who are participating or participated any other clinical trials in latest 30 days will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Study related adverse events | Until week 24

SECONDARY OUTCOMES:
Anti-leukemia response to CART-HER-2 cell infusions | up to 24 weeks

OTHER OUTCOMES:
In vivo existence of CART-HER-2 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Han, Dr., Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Feng K, Liu Y, Guo Y, Qiu J, Wu Z, Dai H, Yang Q, Wang Y, Han W. Phase I study of chimeric antigen receptor modified T cells in treating HER2-positive advanced biliary tract cancers and pancreatic cancers. Protein Cell. 2018 Oct;9(10):838-847. doi: 10.1007/s13238-017-0440-4. Epub 2017 Jul 14. PMID 28710747